CLINICAL TRIAL: NCT00004465
Title: Phase III Randomized Study of SYNSORB Pk in Children With E. Coli-Associated
Brief Title: Phase III Randomized Study of SYNSORB Pk in Children With E. Coli-Associated Hemolytic Uremic Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy at review by DSMB using pre-specified monitoring criteria
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Long Island Jewish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199/13923; LIJMC-96-5-186 (Other: Long Island Jewish Medical Center); R01DK052147 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Hemolytic Uremic Syndrome
Keywords: E. coli infection; bacterial infection; hemolytic uremic syndrome; immunologic disorders and infectious disorders; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Hemolytic-Uremic Syndrome; Escherichia coli Infections; Bacterial Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Urogenital Diseases | interventions — SYNSORB Pk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SYNSORB Pk (Experimental): Oral Shiga toxin-binding agent (500 mg/kg/day)
  Interventions: Drug: SYNSORB Pk
- Placebo (Placebo Comparator): Cornmeal placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYNSORB Pk
  Other Names: Oral Shiga Toxin Binding Agent
  Arms: SYNSORB Pk
Drug: Placebo
  Arms: Placebo

SUMMARY:
OBJECTIVES: I. Determine the effect of SYNSORB Pk therapy on mortality and frequency of severe extrarenal complications observed in children with acute stage E. coli-associated hemolytic uremic syndrome.

II. Determine the effect of SYNSORB Pk therapy on the need for the duration of dialysis in these patients.

III. Determine the effect of SYNSORB Pk therapy on the recovery of renal function and resolution of urinary abnormalities in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are randomized to receive either SYNSORB Pk or placebo.

Patients receive oral SYNSORB Pk or placebo three times daily for 7 days. Patients are followed on days 7, 14, 28, and 60 after discharge from the hospital.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Clinically diagnosed E. coli-associated diarrhea-associated hemolytic uremic syndrome (HUS)
* Diarrheal prodrome within 7 days before onset of disease
* No HUS associated with the following: Hereditary Post-bone marrow transplantation Streptococcus pneumoniae infection
* No prior catastrophic complications

--Patient Characteristics--

* Hematopoietic: Thrombocytopenia less than 140,000/mm3 Fragmented red blood cells
* Renal: Renal involvement (hematuria, proteinuria, or azotemia) No underlying glomerular disease
* Other: HIV negative No pre-existing structural abnormality or dysmotility syndrome of the gastrointestinal tract No inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 1997-07-27 (Actual); Primary Completion 2001-04-14 (Actual); Study Completion 2001-04-14 (Actual)

PRIMARY OUTCOMES:
Time to death or serious extrarenal events | 60 days
Time to dialysis | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, Study Chair — Long Island Jewish Medical Center
Locations (27):
- United States (26):
  - Children's Hospital of Denver, Denver, Colorado
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia Hospital and Clinics, Augusta, Georgia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Children's Hospital at St. Joseph's, Paterson, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Children's Hospital of Buffalo, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Jack D. Weiler Hospital of the Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Bowman Gray School of Medicine, Winston-Salem, North Carolina
  - Ohio State University Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - University of Wisconsin Children's Hospital, Madison, Wisconsin
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trachtman H, Cnaan A, Christen E, Gibbs K, Zhao S, Acheson DW, Weiss R, Kaskel FJ, Spitzer A, Hirschman GH; Investigators of the HUS-SYNSORB Pk Multicenter Clinical Trial. Effect of an oral Shiga toxin-binding agent on diarrhea-associated hemolytic uremic syndrome in children: a randomized controlled trial. JAMA. 2003 Sep 10;290(10):1337-44. doi: 10.1001/jama.290.10.1337. PMID 12966125
- [Derived] Imdad A, Nelson JR, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2025 Apr 25;4(4):CD012997. doi: 10.1002/14651858.CD012997.pub3. PMID 40277027
- [Derived] Imdad A, Mackoff SP, Urciuoli DM, Syed T, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Jul 5;7(7):CD012997. doi: 10.1002/14651858.CD012997.pub2. PMID 34219224